CLINICAL TRIAL: NCT01478386
Title: Randomized Trail to Assess the Effectiveness of an Off-Loading Knee Brace When Combined With Viscosupplementation in the Treatment of Knee Osteoarthritis
Brief Title: Effectiveness of a Knee Brace When Combined With Viscosupplementation in the Treatment of Knee Osteoarthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to poor enrollment
Sponsor: OAD Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Knee OA Treatments
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — orthovisc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Viscosupplementation injections (Other): Control group will receive a series of three viscosupplementation injections into the affected knee
  Interventions: Other: Orthovisc
- Off-loading knee brace (Experimental)
  Interventions: Device: DonJoy HA lite knee brace
- Viscosupplementation and knee brace (Experimental)
  Interventions: Device: Orthovisc injections and DonJoy HA lite knee brace

INTERVENTIONS:
Other: Orthovisc — Subjects will receive a series of three Orthovisc injections into their affected knee
  Arms: Viscosupplementation injections
Device: DonJoy HA lite knee brace — Subjects will be fitted and educated on using the DonJoy HA lite knee brace to treat their affected knee
  Arms: Off-loading knee brace
Device: Orthovisc injections and DonJoy HA lite knee brace — Subjects will receive a series of three Orthovisc injections and be fitted and educated on using a DonJoy HA lite knee brace
  Arms: Viscosupplementation and knee brace

SUMMARY:
Hypothesis: Viscosupplementation when combined with an off-loading knee brace is more effective in treating the symptoms of knee OA then treating with viscosupplementation alone

DETAILED DESCRIPTION:
A randomized prospective study to assess the effectiveness of treating knee osteoarthritis with either a series of three viscosupplementation injections, an off-loading knee brace, or a combination of viscosupplementation and an off-loading knee brace. The viscosupplementation and off-loading knee brace are being used in accordance with their FDA approval. Subjects will be randomized to 1 of 3 treatment groups. The control group will receive a series of weekly (3 consecutive weeks) intra-articular hyaluronic acid injections. The second group will receive a series of weekly (3 consecutive weeks) intra-articular hyaluronic acid injections and an off loading knee brace. The third group will use the off loading knee brace alone. Subjects will complete the WOMAC Osteoarthritis Questionnaire (pain, stiffness, function) and VAS pain scale (measuring pain on movement) at baseline, day 7, day 14, 6 weeks and 3 months. Subjects in group 2 and 3 will be given a brace diary to record compliance.

ELIGIBILITY:
Inclusion criteria:

* Subjects, over the age of 18, with a diagnosis of knee osteoarthritis which is confirmed by radiographs.
* Radiographs will be obtained and patients with mild to moderate knee osteoarthritis will qualify a subject for enrollment.
* Subjects will also have a documented varus deformity.

Exclusion criteria:

* Subjects with severe arthritis as demonstrated by radiographs.
* In addition those subjects with a known or suspected joint infection and subjects who had undergone arthrocentesis and/or intra-articular injection within 3 months of the study will be excluded.
* Female patients who are pregnant or breast feeding will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Reduction in knee pain | 3 months
  The primary outcome measure will be a reduction in knee pain as measured by the VAS pain score. The secondary outcome measure will be an increase in function as measured by the WOMAC Osteoarthritis Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: William R Sterba, MD, Principal Investigator — OAD Orthopaedics
Locations (1):
- OAD Orthopaedics, Warrenville, Illinois, United States